CLINICAL TRIAL: NCT07137936
Title: Comprehensive Cardiac Magnetic Resonance Imaging Evaluation of Myocardial Scar for Predicting Sudden Cardiac Death Post Myocardial Infarction
Brief Title: Cardiac Magnetic Resonance - PROgnostic HEart Scar for Sudden Cardiac Death Prediction StudY
Status: Recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025AZC2006
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Sudden Death, Cardiac; Myocardial Scarring; Myocardial Infarction (MI)
Keywords: sudden cardiac death; myocardial infarction; myocardial scar; Cardiac magnetic resonance imaging
MeSH Terms: conditions — Death, Sudden, Cardiac; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- myocardial infarction patients.: Participants included in this study had previously undergone CMR imaging during the stable phase following their MI as part of their prior clinical care.

SUMMARY:
The purpose of this observational study is to investigate whether myocardial scar characteristics assessed by cardiac magnetic resonance (CMR) can predict the risk of out-of-hospital sudden cardiac death (SCD) after myocardial infarction (MI). It aims to answer two primary questions:

What is the association between CMR-assessed myocardial scar and post-MI SCD? Can we develop an imaging-clinical multimodal risk score for post-MI SCD? Participants included in this study had previously undergone CMR imaging during the stable phase following their MI as part of their prior clinical care. Prognostic data for these participants are collected through clinic visits and telephone follow-up.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) remains a leading cause of mortality post-myocardial infarction (MI). Current risk stratification relying primarily on left ventricular ejection fraction (LVEF ≤35%) for implantable cardioverter-defibrillator (ICD) therapy is inadequate, as many SCD events occur in patients with LVEF >35%. Myocardial scar characteristics assessed by cardiac magnetic resonance (CMR), particularly late gadolinium enhancement (LGE), show promise for improved arrhythmic risk prediction but require robust validation. This study aims to develop and validate a multimodal clinical-CMR risk prediction model integrating comprehensive scar characterization to better identify high-risk post-MI patients who may benefit from ICD therapy, optimizing prevention strategies and resource utilization.

This single-center, ambispective cohort study comprises two phases. Phase 1 (Retrospective): Patients treated for myocardial infarction (MI) at our institution between 2015 and 2025 were screened retrospectively. Those who underwent CMR imaging at least one month post-MI were included. Baseline clinical characteristics and detailed CMR findings were collected. Prognostic data for these patients were retrospectively gathered through January 2026.

Phase 2 (Prospective): Prospective collection of prognostic data for the enrolled cohort will continue from 2026 through 2036. Follow-up will be conducted primarily via clinic visits and telephone interviews at 6-month intervals.

Endpoint Definitions:

Primary Endpoint: Sudden cardiac death (SCD)-equivalent events, encompassing:

SCD events;Aborted SCD events (successful resuscitation from cardiac arrest or ventricular arrhythmia);Appropriate implantable cardioverter-defibrillator (ICD) or cardiac resynchronization therapy defibrillator (CRT-D) therapies for terminating ventricular tachyarrhythmias.

Secondary Endpoints:

Include all-cause mortality, cardiovascular mortality, heart failure rehospitalization, recurrent myocardial infarction, and composite endpoints thereof.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years.
2. Completion of cardiac magnetic resonance (CMR) imaging at Anzhen Hospital during the stable phase (≥1 month) following an acute myocardial infarction (MI).

Exclusion Criteria:

1. Prior implantation of an implantable cardioverter-defibrillator (ICD) or cardiac resynchronization therapy defibrillator (CRT-D) before the index MI.
2. Pre-existing diagnosis of a primary arrhythmia syndrome (e.g., long QT syndrome, Brugada syndrome) before the index MI.
3. Concurrent end-stage disease (e.g., advanced malignancy) directly resulting in an estimated life expectancy of less than one year.
4. History of established non-ischemic cardiomyopathy (e.g., dilated, hypertrophic, or restrictive cardiomyopathy) before the index MI.
5. Significant concomitant valvular heart disease. Status post mechanical heart valve replacement.
6. Patients refuse to be followed up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients with myocardial infarction (MI).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2036-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Sudden cardiac death (SCD)-equivalent events | 10-20 years
  Primary Endpoint: Sudden cardiac death (SCD)-equivalent events, encompassing:
  SCD events: cardiac death occured in a short time period (2 hour of symptom), which were assessed by two separated doctors from the central laboratory.
  Aborted SCD events (successful resuscitation from cardiac arrest or ventricular arrhythmia): patients with ventricular tachycardia, ventricular fibrillation or sudden cardiac arrest who were saved by cardio-pulmonary resuscitation and electric defibrillation.
  Appropriate implantable cardioverter-defibrillator (ICD) or cardiac resynchronization therapy defibrillator (CRT-D) therapies for terminating ventricular tachyarrhythmias: Shock related events were analyzed by two separated experienced electrophysiology doctor,to identify if the shock is delivered by sustained ventricular tachycardia, ventricular fibrillation and sudden cardiac death.

SECONDARY OUTCOMES:
Secondary Outcome | 10-20 years
  Include all-cause mortality, cardiovascular mortality, heart failure rehospitalization, recurrent myocardial infarction, and composite endpoints thereof.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No